CLINICAL TRIAL: NCT06990477
Title: Effect of EIT-guided PEEP On Clinical Outcomes in ARDS Patients With Higher Recuritability: a Pilot Randomized Controlled Trial
Brief Title: Effect of EIT-guided PEEP in ARDS Patients With Higher Recruitability
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, pH.D, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EITVent2
Record Dates: First submitted 2025-05-18; First posted 2025-05-25 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: ARDS (Acute Respiratory Distress Syndrome)
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EIT-guided group (Experimental): Patients will receive PEEP titrated by EIT with a stepwise decrease PEEP trial
  Interventions: Device: EIT-guided PEEP
- low PEEP-FiO2 table group (No Intervention): PEEP will be set according to the low FiO2-PEEP table to keep the oxygenation goals: SpO2 between 88% and 95%, and PaO2 between 55mmHg and 80mmHg.

INTERVENTIONS:
Device: EIT-guided PEEP — PEEP titrated by EIT will be performed with a decremental trial at the enrollment. Right after completing RM, PEEP will be set to 20cmH2O and then reduced in steps of 2cmH2O from 20 to 6 every 2min.
  Arms: EIT-guided group

SUMMARY:
Acute respiratory syndrome distress (ARDS) is a clinical common syndrome with high mortality. Mechanical ventilation (MV) is the cornerstone of management of ARDS but can lead to ventilator-induced lung injury. Positive end-expiratory pressure (PEEP), as one of main component of MV, has been widely used in the clinical practice. However, the PEEP selection is still a difficult problem for moderate to severe ARDS patients. EIT, an imaging tool evaluating the regional ventilation distribution at the bedside, can achieve the individual PEEP selection for all mechanically ventilated patients. Our previous study found that moderate to severe ARDS patients with higher recruitability could benefit from EIT-guided PEEP. This article compared the effect of PEEP titrated guided by EIT with fraction of inspired oxygen (FiO2)-PEEP table on the clinical outcomes in patients with higher recruitability.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years
2. Moderate-to-severe ARDS, defined by the ARDS Definition Task Force in the Berlin definition (partial pressure of arterial oxygen [PaO2]:FiO2 ratio ≤200 mmHg with a PEEP ≥5 cmH2O)
3. RI ratio > 0.5 measured for clinical reasons in the previous 24 hours
4. Diagnosis of ARDS less than 72 hours

Exclusion Criteria:

1. Expected to be mechanically ventilated for less than 48 hours
2. Severe chronic respiratory diseases requiring long-term home oxygen therapy or noninvasive MV
3. Undrained pneumothorax or subcutaneous emphysema
4. Undergoing extracorporeal membrane oxygenation (ECMO) before enrollment
5. Contraindication to the use of EIT (pacemaker, automatic implantable cardioverter defibrillator, and implantable pumps)
6. Severe neuromuscular disease
7. Hemodynamic instability
8. Contraindications to hypercapnia, such as intracranial hypertension or acute coronary syndrome
9. Severe other organs dysfunction with a low expected survival (7 days) or palliative care
10. Solid organ or hematologic tumors with the expected survival time less than 30 days
11. Participating in other clinical trials within 30 days
12. Pregnancy
13. Refusal to sign the informed consent

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2026-01-28 (Actual); Primary Completion 2029-01-19 (Estimated); Study Completion 2029-02-20 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | mortality in Day 28

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Department of Critical Care Medicine, Zhongshan Hospital of Fudan University, Shanghai, China Mainland
  - Department of Critical Care Medicine, Renji Hospital, Shanghai, China Mainland
  - Zhongda Hospital, School of Medicine, Southeast University, Nanjing, Jiangsu